CLINICAL TRIAL: NCT00621465
Title: CTI in the Transition From Hospital to Community
Brief Title: Critical Time Intervention in the Transition From Hospital to Community in People With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01 MH059716,#4640R; R01MH059716 (NIH); DSIR SE-MS
Record Dates: First submitted 2008-02-20; First posted 2008-02-22 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-12

CONDITIONS: Psychotic Disorders
Keywords: Psychosis; Homelessness; Case Management; Severe Mental Illness
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants will receive standard aftercare and community care services.
  Interventions: Behavioral: Usual care
- 2 (Experimental): Participants will receive usual care and the Critical Time Intervention.
  Interventions: Behavioral: Critical Time Intervention (CTI); Behavioral: Usual care

INTERVENTIONS:
Behavioral: Critical Time Intervention (CTI) — CTI is designed specifically to enhance the continuity and focus of care during the transition from psychiatric hospital to community care. CTI does not replace community treatment and support, but instead is meant to complement available services. CTI will provide training in community living skills and in team-managed transfer of caregiving from hospitals to services and supports in the community. Participants will receive CTI for 9 months after hospital discharge.
  Arms: 2
Behavioral: Usual care — Usual care will include the standard aftercare and community care services.

SUMMARY:
This study will evaluate the effectiveness of a psychosocial treatment, Critical Time Intervention, in easing the transition from hospital to community in people with severe mental disorders.

DETAILED DESCRIPTION:
Severe mental illness (SMI) encompasses a wide range of mental disorders and disabilities, but commonly includes disorders that involve symptoms of psychosis. Psychotic symptoms may involve hallucinations, a lost sense of reality, or other distressing symptoms. About 6% of people experiencing psychotic symptoms seek inpatient treatment at a psychiatric hospital. Hospital treatment for a person with SMI often focuses on rapid improvement of negative symptoms and promotion of the necessary skills to successfully return to the community after leaving the hospital. Despite preparation for community integration, the transition from hospital to community remains a difficult time for many people with SMIs, with those affected having an increased chance for suicide, homelessness, and relapse. Critical Time Intervention (CTI), a psychosocial treatment program that aims to restore skills for community living and to assist in seeking service and support in the community, may be more effective than usual care in preventing these adverse outcomes after hospital discharge. This study will compare the effectiveness of CTI versus usual services in preventing homelessness and other adverse outcomes after leaving a psychiatric hospital among people with SMI and psychosis.

Participation in this study will last 18 months. Potential participants will undergo an initial 15- to 30-minute interview that will include questions about current mental, physical, and living conditions; history of psychiatric services; and alcohol and drug use. Eligible participants will then undergo the first full interview, which will include a full review of medical records and will last between 2 and 3 hours. After this interview, participants will be assigned randomly to receive CTI or usual services. For participants assigned to CTI, a CTI specialist will visit participants in the hospital and in their homes and will stay in contact with participants for 9 months after hospital discharge. During visits with the CTI specialist, participants will receive training in community living skills and help finding service and support in the community. Participants assigned to usual services will receive the usual care and community services offered to people recently leaving a psychiatric hospital.

After leaving the hospital, participants in both groups will be asked to participate in 15 follow-up interviews, which will include repeat questions from the 2 initial interviews. Interviews will be conducted once every 6 weeks until 18 months after hospital discharge and will last between 60 and 90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of psychosis
* Homelessness during the 18 months before study entry
* English speaking

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2002-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse outcomes after hospital discharge, particularly homelessness | Measured over 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Herman, DSW, Principal Investigator — NYS Psychiatric Institute
Locations (1):
- Rockland Psychiatric Center, Orangeburg, New York, United States

REFERENCES:
- [Background] Herman D, Conover S, Felix A, Nakagawa A, Mills D. Critical Time Intervention: an empirically supported model for preventing homelessness in high risk groups. J Prim Prev. 2007 Jul;28(3-4):295-312. doi: 10.1007/s10935-007-0099-3. Epub 2007 Jun 1. PMID 17541827